CLINICAL TRIAL: NCT03875248
Title: Arm 1: Optical Blood Pressure Monitoring (OptiBP Mobile App), An Accurate Blood Pressure Measurement Compared to Invasive Blood Pressure Measurement. Arm 2 and Arm 3: Improvement and Validation of the Smartphone Blood Pressure Measurement (OptiBP Mobile App). A Prospective, Method Comparison, Proof of Concept Study in a Swiss Population.
Brief Title: Optical Blood Pressure Monitoring Via Mobile Application, 3 Arms Swiss Clinical Study
Acronym: OPTIBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biospectal (Industry)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Principal Investigator, Patrick Schoettker, Professor, Head of Anaesthesia Unit, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BSP 2018/01
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Intervention Model Description: The arm 1 of the study has been designed as a multicentric prospective pilot study.
  The arm 2 of the study has been designed as a monocentric prospective pilot study.
  The arm 3 of the study has been designed as a monocentric prospective pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1. Blood pressure measurement compared to arterial line (Other): Comparative blood pressure measurement with the investigational device and the invasive reference method (arterial line).
  Interventions: Device: Blood pressure measurement
- Arm 2. Blood pressure measurement compared to manual cuff (Other): Comparative blood pressure measurement in hypertensive patients with the investigational device and the non-invasive reference method (manual cuff).
  Interventions: Device: Blood pressure measurement
- Arm 3. Blood pressure measurement compared to manual cuff (Other): Comparative blood pressure measurement in pregnant women with the investigational device and the non-invasive reference method (manual cuff).
  Interventions: Device: Blood pressure measurement

INTERVENTIONS:
Device: Blood pressure measurement — Measure optically the blood pressure through the use of a smartphone

SUMMARY:
Validation of an existing algorithm designed to estimate blood pressure based on collected optical signals on patients against two reference methods, which are the arterial catheter (arm 1) and the ausculatory sphygmomanometer (arm 2).

DETAILED DESCRIPTION:
The purpose of the study is to compare the blood pressure values measured by a mobile application used with a smartphone and the values measured by reference equipments, which are the arterial line and the ausculatory sphygmomanometer .

In the arm 1 of the study, patients scheduled for general anesthesia at the Centre Hospitalier Universitaire Vaudois (CHUV) and at the Hôpitaux Universitaire de Genève (HUG) will be recruited and their pressure will be measured with both mesurement methods. General anesthesia is known to generate significant variations in blood pressure at the time of induction. During the first minutes of anesthesia, the patient's blood pressure will be measured in parallel with the mobile application and with the reference equipment. After the intervention, the values obtained by the two methods will be compared to confirm the reliability of the data obtained with the mobile application.

In the arm 2, patients scheduled for a medical appointment at the hypertension unit of the Centre Hospitalier Universitaire Vaudois (CHUV) will be recruited. Their pressure will be measured with the mobile application and with the reference equipment at various time points. After the intervention, the values obtained by the two methods will be compared to confirm the reliability of the data obtained with the mobile application.

In the arm 3, patients scheduled for a medical appointment at the maternity unit of the Centre Hospitalier Universitaire Vaudois (CHUV) will be recruited. Their pressure will be measured with the mobile application and with the reference equipment at various time points. After the intervention, the values obtained by the two methods will be compared to confirm the reliability of the data obtained with the mobile application.

ELIGIBILITY:
Arm 1, Inclusion Criteria:

* Informed Consent as documented by signature
* Men or women older than 18 years old
* Good understanding of written and oral speaking used at the centre where the study will be carried out
* American Society of Anesthesiology clinical classification Risk (ASA) Class 1-3
* Scheduled for a general anesthesia
* Necessitating an arterial catheters for the anesthesia and surgery.

Arm 1, Exclusion Criteria:

* Patients that cannot sign informed consent
* Patients in emergency situation, are not legally competent, cannot understand the situation
* ASA Risk class 4
* Dyshythmia like bigeminy, trigeminy, isolated Ventricular Premature Beats (VPB), atrial fibrillation
* Lesion or deficiency on hand, preventing index obstruction of smartphone's camera
* Known contact dermatitis to nickel/chromium

Arm 2, Inclusion Criteria:

* Informed Consent as documented by signature
* Men or women older than 18 years old
* Good understanding of written and oral speaking used at the centre where the study will be carried out

Arm 2,Exclusion Criteria:

* Patients that cannot sign informed consent
* Patients in emergency situation, are not legally competent, cannot understand the situation
* Known or suspected non-compliance (e.g. drug or alcohol abuse, language problems, psychological disorders, dementia)
* Known pregnancy
* Systolic blood pressure difference between two arms >15mmHg or, diastolic blood pressure difference between two arms >10mmHg
* Unstable cardiac condition (myocardial infarction < 1 week, pulmonary embolism, ventricular arrhythmia, decompensated heart failure)
* Dysrhythmia like bigeminy, trigeminy, isolated Ventricular Premature Beats (VPB), atrial fibrillation
* Lesion or deficiency on hand, preventing index obstruction of smartphone's camera
* Known contact dermatitis to nickel/chromium.

Arm 3, Inclusion Criteria:

* Informed Consent as documented by signature
* Pregnant women older than 18 years old
* Good understanding of written and oral speaking used at the centre where the study will be carried out
* Scheduled for a prepartum anesthesia consultation at the hospital maternity unit

Arm 3,Exclusion Criteria:

* Patients that cannot sign informed consent
* Patients in emergency situation, are not legally competent, cannot understand the situation
* Known or suspected non-compliance (e.g. drug or alcohol abuse, language problems, psychological disorders, dementia)
* Systolic blood pressure difference between two arms >15mmHg or, diastolic blood pressure difference between two arms >10mmHg
* Unstable cardiac condition (myocardial infarction < 1 week, pulmonary embolism, ventricular arrhythmia, decompensated heart failure)
* Dysrhythmia like bigeminy, trigeminy, isolated Ventricular Premature Beats (VPB), atrial fibrillation
* Lesion or deficiency on hand, preventing index obstruction of smartphone's camera
* Known contact dermatitis to nickel/chromium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are eligible to take part in the study arm 3. No gender-based eligibility criteria exist for the recruitment of patients in the first and seconf arm of the study.
Enrollment: 350 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2021-06-14 (Estimated)

PRIMARY OUTCOMES:
Confirmation of measurement done with the investigational device | First 20 minutes
  Arm 1: Comparision of values to invasive reference method (arterial line)
Confirmation of measurement done with the investigational device | First 20 minutes
  Arm 2: Comparision of values to non-invasive reference method (ausculatory sphygmomanometer)
Confirmation of measurement done with the investigational device | First 20 minutes
  Arm 3: Comparision of values to non-invasive reference method (ausculatory sphygmomanometer)

SECONDARY OUTCOMES:
Usability assessment | First 20 minutes
  Identification of possible use error in the manipulation of the device and in the performance of the measure
Safety of procedure by assessing inconvenience and adverse events | First 20 minutes
  Safety by assessing inconvenience and adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Hôpital Universitaire de Genève (HUG), Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almeida P, Cuenoud A, Hoang H, Othenin-Girard A, Salhi N, Kothe A, Christen U, Schoettker P. Accuracy of the smartphone blood pressure measurement solution OptiBP to track blood pressure changes in pregnant women. J Hypertens. 2025 Apr 1;43(4):665-672. doi: 10.1097/HJH.0000000000003956. Epub 2025 Feb 7. PMID 39927734
- [Derived] Degott J, Ghajarzadeh-Wurzner A, Hofmann G, Proenca M, Bonnier G, Lemkaddem A, Lemay M, Christen U, Knebel JF, Durgnat V, Burnier M, Wuerzner G, Schoettker P. Smartphone based blood pressure measurement: accuracy of the OptiBP mobile application according to the AAMI/ESH/ISO universal validation protocol. Blood Press Monit. 2021 Dec 1;26(6):441-448. doi: 10.1097/MBP.0000000000000556. PMID 34139747